CLINICAL TRIAL: NCT02690376
Title: An Observer Blinded Comparison of Magnetically Assisted Capsule Endoscopy and Conventional Upper Gastrointestinal Endoscopy in Upper GI Bleeding
Brief Title: An Observer Blinded Comparison of MACE and Conventional Upper Gastrointestinal Endoscopy in Upper GI Bleeding
Acronym: MACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: IntroMedic USA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH19107
Record Dates: First submitted 2016-02-10; First posted 2016-02-24 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Gastrointestinal Diseases
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magnetic Assisted Capsule Endoscopy (Other): There is only one arm and its does not reach criteria for other options
  Interventions: Device: Magnetic Assisted Capsule Endoscopy

INTERVENTIONS:
Device: Magnetic Assisted Capsule Endoscopy — Swallowed magnetic capsule for endoscopy purposes
  Other Names: MACE

SUMMARY:
Gastroscopy (OGD) is a useful test for investigating a variety of suspected upper GI disorders. But it is uncomfortable for patients and incurs the risk of intubation and sedation, plus a large proportion of procedures reveal insignificant or no pathology. Capsule endoscopy (CE) is the investigation of choice for diseases of the small bowel. It is safe, non-invasive and well-tolerated. The use of CE is traditionally restricted to the small bowel, although newer capsules to image the oesophagus and colon are currently in use. Previous capsules have failed to adequately image the stomach due to its' large volume and rugal folds. Recently a magnetic capsule and handheld magnet has been developed (Mirocam Navi, Intromedic Ltd, Seoul, Korea) to enable an element of manoeuvrability of the capsule. This is unnecessary in the small bowel where the capsule is propelled along its' tubular structure by peristalsis, but in the capacious stomach this may allow the capsule to be steered to examine all areas of the stomach. We have already conducted two feasibility studies in porcine models with promising results and a trial has already evaluated the equipment to steer the small bowel capsule through the stomach into the duodenum. An ongoing study is comparing the ability of this technique to examine the stomach against conventional OGD, in patients with recurrent iron deficiency anaemia. The next stop would be to compare the two modalities under other different conditions.

We wish to undertake a prospective single blind controlled trial comparing magnetically assisted capsule examination to conventional OGD in diagnosing upper gastrointestinal pathology in patients with gastrointestinal bleeding.

DETAILED DESCRIPTION:
Intubational endoscopy is uncomfortable for patients and incurs the risks of bleeding, perforation and sedation related complications. Gastroscopy is the 'gold-standard' investigation to identify upper gastrointestinal pathology but is poorly tolerated by patients. Moreover a large proportion of gastroscopies are normal or reveal insignificant pathology and despite efforts to produce pre-procedure scoring systems to grade the appropriateness of the procedure, correlation with diagnostic yield is poor. Capsule endoscopy is very well tolerated but is traditionally reserved for examination of the small bowel since it cannot be manipulated to view all areas of the capacious stomach. A capsule which could overcome this and be steered to examine all areas of the mucosal surface of the stomach as an alternative to intubational endoscopy would be advantageous to patients. Mirocam Navi (MC1000-WM, Intromedic Ltd, Seoul, Korea) is a small bowel capsule endoscope with an inclusion of magnetic material. Available accessories include a handheld magnet with which to gain some control over the capsule in the upper gastrointestinal tract. The capsule is CE marked (CE0120) with the handheld magnet classed as an accessory. In order to assess the feasibility of our hypothesis we conducted a study in an ex vivo porcine stomach model, commonly used for endoscopy training purposes. Different coloured/shaped beads were sewn into each major location of the stomach (cardia, fundus, greater and lesser curve, anterior and posterior wall, antrum and D1). The stomach was distended with 1000mls of water. Endoscopy was performed according to a set protocol. All stomach tags were identified in 87.2% (41/47) of examinations.

This was followed by a double blind, randomised controlled trial comparing magnetically assisted capsule endoscopy (MACE) with conventional upper gastrointestinal endoscopy to detect coloured beads in a porcine stomach model. Gastroscopy correctly identified 88% (79/90) beads, MACE correctly identified 89% (80/90) beads and thus is noninferior to gastroscopy in this setting (95% CI 82.76%-95.24%). Mean examination times for gastroscopy and MACE were 3.34 minutes and 9.90 minutes respectively. Clearly there are significant differences between a porcine model and live human stomach. However, these studies provide proof of the principle that a small bowel capsule endoscope can be manipulated to make targeted movements within the stomach. We now also have one completed human trial assessing whether the magnetic controller can be utilised to manipulate the small bowel capsule through the stomach into the duodenum to improve the completion rate of small bowel capsule examinations. Another trial is also near completion comparing the diagnostic ability ,within the stomach, of MACE compared to conventional gastroscopy in the context of recurrent iron deficiency anaemia.

In order to develop the protocol for our study, discussions were made with other health professionals (consultants, specialist nurses and ward nurses) who are involved in performing or reporting gastroscopy and small bowel capsule endoscopy examinations outside of the research team. Feedback was used to modify the study protocol so it could be as patient and user friendly as possible without compromising the overall aim to answer the research question.

Additionally the protocol has been externally peer reviewed and subsequent modifications made.

From our porcine and two human trials it is clear that to obtain reasonable views of the stomach to be able to guide the capsule the stomach needs to be distended. In our porcine study we achieved good results with 1000mls of water. We felt that this would be an acceptable amount for a patient to drink prior to magnetically assisted capsule endoscopy, and the two human trials we have completed to date have proven excellent tolerance to this volume of water.

RECRUITMENT Patients will be offered information about the trial at the time of their initial clinical encounter in the outpatient clinic. Written information is provided at this stage and will be followed by confirmation of consent on the day of, but prior to, the procedure. The research team will be available when the patient attends for their procedures to answer any questions or concerns. Additionally a contact telephone number for the research team is provided on the patient information sheet for any other concerns or queries.

INCLUSION/EXCLUSION We have made every effort to enable the study to be open to a wide range of patients however we have currently limited the study to patients with upper gastrointestinal bleeding to allow the highest possibility for pathology detection for either endoscopic modality and hence facilitate comparison of diagnostic ability. Specific considerations have been made to ensure that patients will be excluded from the study if there is to be any delay/interference to the standard management of upper gastroinstinal bleeding.

CONSENT All participants will be consented as per the study consent form. All members of the research team are formally trained in consent procedures and assessment of capacity. Any participant without capacity to consent will not be included in the trial. The principal investigator is trained in the ethical principles underpinning informed consent and is bound to these principles as part of good medical practice.

RISKS/BURDENS/BENEFITS The participant is subject to the risk of the procedures of gastroscopy and small bowel capsule endoscopy itself. Bleeding and perforation are the major risks of undergoing a gastroscopy and occur in 0.02% of procedures. There is also a risk of sedation related complications if the patient chooses this option. The main risk of SBCE is retention of the capsule, occurring in up to 2% of examinations. Since the participant is undergoing these procedures as part of their medical investigation these risks are discussed when the patient is offered the investigations at the time of booking, they are also formally consented by a trained individual when they attend for the procedure. Participants are not felt to be at any additional risk by undergoing magnetically steerable capsule examination of the stomach.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over
* Patients presenting with haematemesis (fresh blood or coffee grounds) and/or malaena within the previous 48 hours, who require a gastroscopy as part of their diagnostic investigations

Exclusion Criteria:

* Patients under the age of 18 years or over the age of 80 years.
* Patients who have a suspected UGIB and haemodynamic instability, i.e. hypotension (systolic blood pressure <100mmHg) and tachycardia (>100 bpm), requiring urgent resuscitation
* Pre-endoscopy Rockall score >4 (patients with a lower pre-endoscopy Rockall score but haemodynamically unstable will still be excluded)
* Active vomiting or haematemesis
* Patients with a permanent pacemaker, implantable cardioverter-defibrillator or REVEAL device
* Patients with any electronic/magnetic/mechanically controlled devices e.g. sacral nerve stimulators, bladder stimulators
* Patients with dysphagia, odynophagia or known swallowing disorder
* Patients with known Zenker's diverticulum
* Patients with suspected bowel obstruction or bowel perforation
* Patients with prior bowel obstruction
* Patients with gastroparesis or known gastric outlet obstruction
* Patients with known Crohn's disease
* Patients with a history of GI tract surgery (Billroth I, Billroth II, Oesophagectomy, gastrectomy or bariatric procedure)
* Patients that are pregnant or lactating
* Patients with altered mental status that would limit their ability to swallow
* Patients with allergy to conscious sedation or metoclopramide
* Patients unwilling to swallow the capsule
* Patients unwilling to undergo a possible abdominal XR if suspected capsule retention occurs
* Patients with known dementia affecting ability to consent
* Patients who are unable to understand or speak English
* Patients unable to provide written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of pathology of MACE compared to gastroscopy. | Baseline - one visit only

SECONDARY OUTCOMES:
Mucosal visualisation of the oesophagus and major areas of the stomach during MACE. | Baseline - one visit only
Determine the number of patients with small bowel bleeding | Baseline - one visit only
Tolerability of MACE compared to gastroscopy | Baseline - one visit only
Duration of MACE compared to gastroscopy | Baseline - one visit only
Determine if MACE can be used to avoid unnecessary OGD or hospital admission | Baseline - one visit only

CONTACTS AND LOCATIONS:
Overall Officials: Mark McAlindon, Dr, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Royal Hallamshire Hospital, Sheffield, South Yorkshire
  - Sheffield Teaching Hospitals FT Trust, Sheffield, South Yorkshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ching HL, Hale MF, Sidhu R, Beg S, Ragunath K, McAlindon ME. Magnetically assisted capsule endoscopy in suspected acute upper GI bleeding versus esophagogastroduodenoscopy in detecting focal lesions. Gastrointest Endosc. 2019 Sep;90(3):430-439. doi: 10.1016/j.gie.2019.04.248. Epub 2019 May 10. PMID 31082392